CLINICAL TRIAL: NCT06487975
Title: Effects of Bacillus Subtilis on Blood and Gut Biomarkers in Parkinson's Disease
Brief Title: Bacillus Subtilis in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Helse Stavanger HF (Other Government); ADM Protexin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 22/WS/0100
Record Dates: First submitted 2024-03-27; First posted 2024-07-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: probiotic; microbiome
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus Subtilis (Experimental): Bacillus Subtilis 1 capsule once daily in the morning (consisting of 10x10^9 Colony Forming Units)
  Interventions: Dietary Supplement: Bacillus Subtilis
- Placebo (Placebo Comparator): 1 visually identical placebo capsule once daily in the morning using the same carrier (microcrystalline cellulose) as the active (but not containing Bacillus Subtilis)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus Subtilis — Bacillus Subtilis 1 capsule once daily in the morning (consisting of 10x10^9 Colony Forming Units)
  Arms: Bacillus Subtilis
Other: Placebo — 1 visually identical placebo capsule once daily in the morning using the same carrier (microcrystalline cellulose) as the active (but not containing Bacillus Subtilis)
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate whether the administration of Bacillus Subtilis influences gut and blood biomarkers relevant to the proposed mechanism(s) of action, as well as being acceptable as a regular supplement for people with Parkinson's disease.

DETAILED DESCRIPTION:
Following informed consent, participants will undergo screening. If eligible, they will be invited to attend a baseline visit (week 0) to complete clinical assessments and provide a faecal and blood sample before starting their assigned intervention. Each participant will be randomised 1:1 to visually identical capsules containing either Bacillus Subtilis or placebo to be taken for 24 weeks. Telephone follow-up will be performed at week 8 to ensure compliance and answer any participant questions. Repeat clinical assessments and faecal/blood sample collection will take place at weeks 24 (treatment end date) and 36 (to assess longevity of biomarker changes after the intervention has stopped). Faecal samples will be collected at home within seven days prior to the clinic visits and brought to the appointment. Microbiota composition in faecal samples and blood biomarkers will be analysed in participant samples. Motor and non-motor symptom rating scales will also be administered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Able to provide written informed consent
* Over 50 years old
* Motor symptom duration over 12 months
* Stable dopaminergic medication regime for at least 3 months

Exclusion Criteria:

* Use of probiotic supplements and probiotic-fortified foods (such as probiotic drinks and yoghurts) within past 3 months
* Use of antibiotics within past 3 months
* Previous gastrointestinal surgery or chronic organic bowel disorder
* History of clinically significant motor fluctuations
* History of postural instability or falls
* Current smoker
* Known or suspected allergy to probiotics
* Regular use of antacids, proton pump inhibitors, laxatives or anti-diarrheal drugs
* Use of hypoglycaemic or diabetes drugs
* Participation in clinical trial of investigational medicinal product within past 3 months
* Co-morbidities or other factors that, in the opinion of the investigator, make the patient unlikely to comply with study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of Bacillus Subtilis on gut microbiome | 24 weeks
  Changes in presence and abundance of Bacillus Subtilis and other bacteria in faeces following probiotic administration versus placebo. Non-parametric tests (such as Wilcoxon signed-rank test and permutational multivariate analysis of variance) will be used for alpha and beta diversity analyses, and to identify genera that have significantly changed in abundance.
To assess the effects of Bacillus Subtilis on blood biomarkers (sphingolipid profile) | 24 weeks
  Changes in sphingolipids following Bacillus Subtilis administration versus placebo measured using liquid chromatography-mass spectrometry
To assess the effects of Bacillus Subtilis on blood biomarkers (pro-inflammatory cytokines) | 24 weeks
  Changes in pro-inflammatory cytokines following Bacillus Subtilis administration versus placebo measured using V-PLEX Proinflammatory Panel 1 Human Kit
To assess the effects of Bacillus Subtilis on blood biomarkers (neurofilament light chain) | 24 weeks
  Changes in neurofilament light chain following Bacillus Subtilis administration versus placebo measured using Single Molecule Array assay
To assess the effects of Bacillus Subtilis on blood biomarkers (alpha-synuclein species) | 24 weeks
  Changes in alpha synuclein species following Bacillus Subtilis administration versus placebo measured using α-syn real-time quaking-induced conversion assays
To assess the effects of Bacillus Subtilis on blood biomarkers (lipid profile) | 24 weeks
  Changes in cholesterols/triglycerides following Bacillus Subtilis administration versus placebo
To assess the effects of Bacillus Subtilis on blood biomarkers (fasting glucose) | 24 weeks
  Changes in fasting glucose following Bacillus Subtilis administration versus placebo
To assess the effects of Bacillus Subtilis on blood biomarkers (haemoglobin A1C) | 24 weeks
  Changes in haemoglobin A1C following Bacillus Subtilis administration versus placebo
To evaluate the acceptability of Bacillus Subtilis administration in PD patients | 24 weeks
  Descriptive analysis of custom-designed Acceptability Questionnaire which includes four questions on number of missed doses, ease of swallowing, daily dosing schedule, and any other barriers to tablet compliance.

SECONDARY OUTCOMES:
To evaluate the correlation between changes in gut and blood biomarkers following B. subtilis administration and motor/non-motor symptoms | 24 weeks
  Correlation between Primary Objectives 1 and 2 and motor/non-motor symptoms: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Movement Disorder Society Non-Motor Rating Scale (MDS-NMS), Montreal Cognitive Assessment (MoCA) and Parkinson's Disease Questionnaire (PDQ-39)

CONTACTS AND LOCATIONS:
Overall Officials: David P Breen, MBChB, Study Chair — NHS Lothian
Locations (2):
- Norwegian Centre for Movement Disorders, Stavanger University Hospital, Stavanger, Norway
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No